CLINICAL TRIAL: NCT00778921
Title: A Randomized, Eight Week Double-blind, Parallel-group, Multicenter Study to Evaluate the Efficacy and Safety of the Combination of Aliskiren / Amlodipine (150/10 mg and 300/10 mg) in Comparison With Amlodipine 10 mg in Patients With Essential Hypertension Not Adequately Responsive to Amlodipine 10 mg Monotherapy
Brief Title: Study to Evaluate the Efficacy and Safety of Combination Aliskiren/Amlodipine in Patients With Hypertension Not Adequately Responding to Amlodipine Alone
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Study Director, Novartis Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSPA100A2304
Record Dates: First submitted 2008-10-23; First posted 2008-10-24 (Estimated); Results first posted 2011-03-23 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2011-02

CONDITIONS: Hypertension
Keywords: Aliskiren; Amlodipine; Non-responder to Amlodipine
MeSH Terms: conditions — Hypertension | interventions — Amlodipine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Amlodipine 10 mg (Experimental): Amlodipine 10 mg
  Interventions: Drug: Amlodipine 10 mg
- Aliskiren/Amlodipine 150/10 mg (Experimental): Aliskiren/Amlodipine 150/10 mg
  Interventions: Drug: Amlodipine 10 mg; Drug: Aliskiren 150
- Aliskiren/Amlodipine 300/10 mg (Experimental): Aliskiren/Amlodipine 300/10 mg
  Interventions: Drug: Amlodipine 10 mg; Drug: Amlodipine 300

INTERVENTIONS:
Drug: Amlodipine 10 mg — Amlodipine 10 mg
Drug: Aliskiren 150 — Aliskiren/Amlodipine 150/10 mg
  Arms: Aliskiren/Amlodipine 150/10 mg
Drug: Amlodipine 300 — Aliskiren/Amlodipine 300/10 mg
  Arms: Aliskiren/Amlodipine 300/10 mg

SUMMARY:
This study will assess the safety and efficacy of combination aliskiren/amlodipine in patients with hypertension not adequately controlled with amlodipine alone.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed patients or patients who have not been treated for hypertension within the 4 weeks prior to Visit 1 must have a msDBP ≥ 95 mmHg and < 110 mmHg at Visits 1 and 2
* Patients who have been treated for hypertension within the 4 weeks prior to Visit 1 must have a msDBP ≥ 90 mmHg and < 110 mmHg at Visit 2
* All patients must have a msDBP ≥ 90 mmHg and < 110 mmHg at Visit 5 (randomization)

Exclusion Criteria:

* Severe hypertension
* Pregnant or nursing (lactating) women
* Pre-menopausal women not taking accepted form of birth control
* Serum potassium ≥ 5.3 mEq/L (mmol/L) at Visit 1
* History of cardiovascular conditions
* Uncontrolled Type 1 or Type 2 diabetes mellitus
* Hypersensitivity to renin inhibitors, calcium channel blockers, or to drugs with similar chemical structures

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 847 (Actual)
Dates: Start 2008-10; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Chair — N
Locations (7):
- Investigative Site, Buenos Aires, Argentina
- Investigative Site, Berlin, Germany
- Investigative Site, Oslo, Norway
- Investigative Site, Warsaw, Poland
- Investigative Site, Bratislava, Slovakia
- Investigative Site, Stockholm, Sweden
- Investigative Site, Ankara, Turkey (Türkiye)

REFERENCES:
- [Derived] Pfeiffer D, Rennie N, Papst CC, Zhang J. Efficacy and tolerability of aliskiren/amlodipine single-pill combinations in patients who did not respond fully to amlodipine monotherapy yen. Curr Vasc Pharmacol. 2012 Nov;10(6):773-80. doi: 10.2174/157016112803520945. PMID 22303911

RESULTS

PARTICIPANT FLOW:
Groups:
- Aliskiren/Amlodipine 300/10 mg: Oral tablets of combination aliskiren/amlodipine 300/10 mg taken once daily with water in the morning
- Aliskiren/Amlodipine 150/10 mg: Oral tablets of combination aliskiren/amlodipine 150/10 mg taken once daily with water in the morning
- Amlodipine 10 mg: Oral capsules of amlodipine 10 mg taken once daily with water in the morning
Period: Overall Study
Arm/Group | Aliskiren/Amlodipine 300/10 mg | Aliskiren/Amlodipine 150/10 mg | Amlodipine 10 mg
Started | 279 | 285 | 283
Completed | 261 | 266 | 255
Not Completed | 18 | 19 | 28
Not completed — Adverse Event | 9 | 10 | 14
Not completed — Abnormal Laboratory Value(s) | 1 | 0 | 0
Not completed — Abnormal Test Procedure Result(s) | 0 | 0 | 2
Not completed — Unsatisfactory therapeutic response | 1 | 1 | 1
Not completed — Patient No Longer Requires Study Drug | 0 | 1 | 0
Not completed — Patient withdrew request | 3 | 1 | 6
Not completed — Lost to Follow-up | 0 | 2 | 1
Not completed — Administrative Problems | 1 | 2 | 0
Not completed — Protocol Violation | 3 | 0 | 2
Not completed — Not treated | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aliskiren/Amlodipine 300/10 mg | Aliskiren/Amlodipine 150/10 mg | Amlodipine 10 mg | Total
Number analyzed (Participants) | 279 | 285 | 283 | 847
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.2 (10.19) | 54.4 (10.70) | 54.3 (10.92) | 54.6 (10.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 116 | 113 | 99 | 328
  Male | 163 | 172 | 184 | 519

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Sitting Diastolic Blood Pressure (msDBP) From Baseline to End of Study
Time Frame: Baseline and Week 8
Population: full analysis set
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Aliskiren/Amlodipine 300/10 mg | Aliskiren/Amlodipine 150/10 mg | Amlodipine 10 mg
Number analyzed (Participants) | 277 | 281 | 279
mm Hg | -10.99 (0.462) | -8.95 (0.460) | -7.23 (0.459)

2. Secondary Outcome: Change in Mean Sitting Systolic Blood Pressure (msSBP) From Baseline to End of Study
Time Frame: Baseline and Week 8
Population: full analysis set
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Aliskiren/Amlodipine 300/10 mg | Aliskiren/Amlodipine 150/10 mg | Amlodipine 10 mg
Number analyzed (Participants) | 277 | 281 | 279
mm Hg | -14.42 (0.684) | -11.01 (0.681) | -8.20 (0.680)

3. Secondary Outcome: Number of Patients With Any Adverse Event and/or Serious Adverse Event in the Double-blind Period by Treatment Group
Time Frame: 8 weeks
Population: Analysis: Intention to Treat (ITT) Imputation Technique: Last Observation Carried Forward (LOCF)
Measure: Number; unit: Participants
Arm/Group | Aliskiren/Amlodipine 300/10 mg | Aliskiren/Amlodipine 150/10 mg | Amlodipine 10 mg
Number analyzed (Participants) | 279 | 283 | 281
Participants | 87 | 99 | 92

4. Secondary Outcome: Biomarker Assessment at Visit 2 (Single Blind Run in), Visit 5 (Randomization), and Visit 9 (EOS)
Time Frame: 12 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Groups:
- Aliskiren 300mg/ Amlodipine 10mg: Aliskiren 300mg/ Amlodipine 10mg
- Aliskiren 150mg/ Amlodipine 10mg: Aliskiren 150mg/ Amlodipine 10mg
- Amlodipine 10mg: Amlodipine 10mg
Arm/Group | Aliskiren 300mg/ Amlodipine 10mg | Aliskiren 150mg/ Amlodipine 10mg | Amlodipine 10mg
Serious Adverse Events (participants affected / at risk) | 4/279 | 1/283 | 0/281
Other Adverse Events (participants affected / at risk) | 31/279 | 35/283 | 40/281
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aliskiren 300mg/ Amlodipine 10mg (N=279) | Aliskiren 150mg/ Amlodipine 10mg (N=283) | Amlodipine 10mg (N=281)
Lymphoid tissue hyperplasia (Blood and lymphatic system disorders) | 1 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Renal artery stenosis (Renal and urinary disorders) | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aliskiren 300mg/ Amlodipine 10mg (N=279) | Aliskiren 150mg/ Amlodipine 10mg (N=283) | Amlodipine 10mg (N=281)
Oedema peripheral (General disorders) | 15 | 23 | 25
Nasopharyngitis (Infections and infestations) | 16 | 15 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.